CLINICAL TRIAL: NCT01169714
Title: An Investigator And Subject-Blind Phase 1 Study To Characterize The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Doses Of PF-04995274 In Healthy Adult And Healthy Elderly Subjects
Brief Title: A Study To Observe Safety And Blood Concentrations Of PF-04995274 During And Following the Administration of Multiple Doses Of PF-04995274 In Healthy Adult And Healthy Elderly Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B1661003
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: multiple dose; healthy volunteer; healthy elderly volunteer; safety; pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dosing Healthy Adult (Experimental): Ascending Doses in Healthy Adult Volunteers
  Interventions: Drug: 0.1 mg PF-04995274; Drug: 1 mg PF-04995274; Drug: 10 mg PF-04995274; Drug: 15 mg PF-04995274
- Dosing Healthy Elderly (Experimental): Dosing in Healthy Elderly volunteers
  Interventions: Drug: 1.0 mg PF-04995274; Drug: 15 mg PF-04995274

INTERVENTIONS:
Drug: 0.1 mg PF-04995274 — 0.1 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Adult
Drug: 1 mg PF-04995274 — 1 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Adult
Drug: 10 mg PF-04995274 — 10 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Adult
Drug: 15 mg PF-04995274 — 15 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Adult
Drug: 1.0 mg PF-04995274 — 1.0 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Elderly
Drug: 15 mg PF-04995274 — 15 mg PF-04995274, qd, for 14 days or placebo
  Arms: Dosing Healthy Elderly

SUMMARY:
This study is designed to observe the safety and blood concentrations of PF-04995274 during and following the administration of multiple doses of PF-04995274 for a duration of 14 days, in healthy adult and healthy elderly.

DETAILED DESCRIPTION:
To examine the safety and pharmacokinetics of PF-04995274 in healthy adult and healthy elderly subjects after multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy adult volunteers: healthy male and/or female subjects of non child bearing potential between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests.)
* For Healthy Elderly volunteers: healthy male and/or female subjects of non child bearing potential between the ages of 65 and 85 years, inclusive. Subjects must be in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12 lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease (eg, controlled hypertension, non-insulin dependent diabetes, osteoarthritis) may be enrolled if deemed medically prudent by the investigator. In order to ensure an age range relevant to the Alzheimer's Disease (AD) population, no more than 30% of subjects enrolled in any cohort may be less than 70 years of age.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints (Adverse events, Change from baseline in vital signs, Change from baseline in triplicate ECGs, Clinical safety laboratory, Clinical examinations, Digit Symbol Substitution Test (DSST)) | Day 0 to Day 28
Pharmacokinetic endpoints Plasma concentration of PF 04995274 over time (eg, AUC, Cmax, Tmax, t1/2), Plasma concentration of PF 05082547 over time (eg, AUC, Cmax, Tmax, t1/2). | Day 0 to Day 28
Pharmacodynamic endpoint Aldosterone concentration in healthy adult subjects. | Day 0 to Day 14

SECONDARY OUTCOMES:
No secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1661003&StudyName=A%20Study%20To%20Observe%20Safety%20And%20Blood%20Concentrations%20Of%20PF-04995274%20During%20And%20Following%20the%20Administration%20of%20Multiple%20Doses%20Of%20PF-049952